CLINICAL TRIAL: NCT06488560
Title: The Impact of Commercial Blenderized Formula on Caloric Needs, Gastrointestinal Symptoms, and Gut Microbiome in Children With Cerebral Palsy: A Single Center Randomized Open Label Clinical Trial
Brief Title: The Impact of Commercial Blenderized Formula on Caloric Needs, Gastrointestinal Symptoms, and Gut Microbiome in Children With Cerebral Palsy (CP)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Fernando Navarro, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HSC-MS-24-0047
Record Dates: First submitted 2024-05-07; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Cerebral Palsy
Keywords: Blenderized tube feeds (BTF); commercial blenderized tube feed (CBTF); Commercial formula
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- commercial blenderized tube feed (CBTF) (Experimental)
  Interventions: Dietary Supplement: commercial blenderized tube feed (CBTF)
- commercial formulas (CF) (Active Comparator)
  Interventions: Dietary Supplement: commercial formulas (CF)

INTERVENTIONS:
Dietary Supplement: commercial blenderized tube feed (CBTF) — Based on assessment by a dietician the participant will be fed the commercial blenderized formula to meet their caloric needs
  Arms: commercial blenderized tube feed (CBTF)
Dietary Supplement: commercial formulas (CF) — Participant will be fed the commercial formula to meet their caloric needs per standard of care
  Arms: commercial formulas (CF)

SUMMARY:
The purpose of this study is to compare the Pediatric Quality of Life Inventory Gastrointestinal Symptoms Scale Gastrointestinal Symptoms Scale (GI-PedsQL) differences , to assess the differences in stool microbiome and stool metabolomics , to assess differences in salivary cytokine profile , to assess differences in weight change , to compare the use of antacid medications and to compare the use of laxative medications in patients on commercial formulas (CF) versus commercial blenderized tube feed (CBTF).

ELIGIBILITY:
Inclusion Criteria:

* Patients with CP receiving >75% of total daily caloric requirements from commercial formulas (CF) via a gastrostomy tube 12french or greater
* Patients' insurance covers a CBTF
* Diagnosis of cerebral palsy

Exclusion Criteria:

* Receiving enteral nutrition by transpyloric feeds or jejunal tube.
* Receiving <75% of total daily energy requirements from a commercial formula
* Weight or weight for length or body mass index less than the 5th percentile for age or greater than the 85th% percentile for age when plotted on the cerebral palsy growth chart
* Rapidly progressive neurodegenerative disease diagnosis
* Use of monomeric formulas

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life as assessed by the Pediatric QoL Inventory of GI Symptom Scale. | Baseline, end of study (2 months after baseline)
  This is a 74 item questionnaire and each is scored from 0 (never) to 4 (almost always), higher score indicating worse outcome.

SECONDARY OUTCOMES:
Change in fecal samples for microbiome analysis (identity, composition, and relative abundance of bacterial taxa in stool specimens) | Baseline, end of study (2 months after baseline)
Change in stool metabolomic profile | Baseline, end of study (2 months after baseline)
  Mass spectrometry will be used to assess the following metabolites: amino acids, methylated metabolites, bile acids, and nucleotides.
Change in salivary cytokine profile | Baseline, end of study (2 months after baseline)
  Gene expression of the following salivary inflammatory cytokines will be assessed: interleukin-8 (IL-8), toll-like receptor 8 (TLR8), interleukin-26 (IL-26), interleukin-22 (IL-22), C-C motif chemokine receptor type 1 (CCR1), Caspase 2 (CASP2), toll-like receptor 8 (TLR8), and Intercellular adhesion molecule 3 (ICAM3).
Change in stool caliber using the Bristol stool scale | Baseline, end of study (2 months after baseline)
  The Bristol stool scale categorizes stool into one of 7 types, as follows. Types 1 and 2 indicate constipation, with 3 and 4 being the ideal stools as they are easy to defecate while not containing excess liquid, and 6 and 7 indicate diarrhea.
  Type 1: Separate hard lumps, like nuts (difficult to pass) Type 2: Sausage-shaped, but lumpy Type 3: Like a sausage but with cracks on its surface Type 4: Like a sausage or snake, smooth and soft (average stool) Type 5: Soft blobs with clear cut edges Type 6: Fluffy pieces with ragged edges, a mushy stool (diarrhea) Type 7: Watery, no solid pieces, entirely liquid (diarrhea)
Number of participants who needed to add or remove antacid or laxative medications from their bowel regimen | Baseline, end of study (2 months after baseline)
  Medications in the bowel regimen include antacids and laxatives.
Number of participants who had dose adjustments to their antacid or laxative medications | Baseline, end of study (2 months after baseline)
Change in weight | Baseline, end of study (2 months after baseline)
Change in weight percentile | Baseline, end of study (2 months after baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Navarro, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No